CLINICAL TRIAL: NCT05166265
Title: A Prospective, Multi-center, Single-arm, Clinical Investigation of the Safety and Performance of the Sentio System in Users With Mixed/Conductive Hearing Losses and Single Sided Deafness
Brief Title: Clinical Investigation Study of Safety and Performance of the Sentio System.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC101; CIV-21-07-037287 (Other: EUDAMED); CI/2021/0043/GB (Other: MHRA)
Record Dates: First submitted 2021-12-08; First posted 2021-12-21 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Hearing Loss, Conductive; Hearing Loss, Mixed; Hearing Loss, Unilateral
Keywords: Hearing Loss; Conductive; Mixed; Single-sided; Deafness
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Hearing Loss, Unilateral; Hearing Loss; Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sentio system (Experimental): Prospective, open label, single-arm multi-centre investigation following clinical practice for bone conduction devices.
  Interventions: Device: Active transcutaneous bone conduction hearing system

INTERVENTIONS:
Device: Active transcutaneous bone conduction hearing system — The Sentio system consists of the Sentio 1 sound processor (SP) and Sentio Ti implant with fixation band and screws.
  Other Names: Sentio system

SUMMARY:
Prospective, open label, single-arm, multi-centre investigation, designed to follow clinical practice for Sentio bone conduction devices in 50 subjects, during 10 clinical visits, and 24 months follow-up.

DETAILED DESCRIPTION:
The investigation is a 24-months multinational, multicentre, prospective, open label, single arm investigation on the Sentio system. The purpose of this investigation is to evaluate safety and performance three months after implantation of the new Sentio system. In addition, safety will be analysed six months after implantation, and long-term safety and performance will be evaluated over a 24-month follow-up period. The endpoints chosen, together with applicable measurements, are commonly used, both in the clinical setting as well as in bone anchored hearing research as shown in the scientific literature covering this area. That is, the primary objectives of this study is to demonstrate that the Sentio system improves hearing and speech recognition on the implanted ear. Secondary objectives includes investigation of hearing improvement, speech intelligibility, patient satisfaction, and quality of life. The study also aims to evaluate the safety profile of the Sentio system in terms of the occurrence of adverse events and serious adverse events related to the device.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Adult subjects (18 years or older)
3. Subjects with 3.1. conductive or mixed hearing losses with pure tone average (PTA) bone conduction (BC) threshold (measured at 0.5, 1, 2 and 3 kHz) of the indicated ear better than or equal to 45 dB HL.

   3.2. OR subjects who have a profound sensorineural hearing loss in one ear and normal hearing in the opposite ear (i.e. SSD). The pure tone average (PTA) air conduction (AC) threshold of the hearing ear should then be better than or equal to 20 dB HL (measured at 0.5, 1, 2 and 3 kHz) 3.3. OR subjects who are indicated for an air-conduction contralateral routing of signals (ACCROS) hearing aid, but who for some reason cannot or will not use an AC CROS.
4. Fluent in local language
5. Subjects who have the ability and are willing to follow investigational procedures/requirements, e.g. to complete quality of life scales.

Exclusion Criteria:

1. Inability to undergo general or local anesthesia
2. Prior implantation with percutaneous device or middle ear implant on the side to be implanted
3. Known medical conditions that contraindicate undergoing surgery as judged by the investigator
4. Untreated ongoing middle ear infection at the time of surgery
5. Known insufficient bone quality/quantity/depth or skull size (scull abnormalities) for implantation of a Sentio Ti Implant
6. Known or suspected contact allergy to silicone or other material used in the Sentio system.
7. Known condition that could jeopardize wound healing and skin condition e.g. uncontrolled diabetes over time as judged by the investigator.
8. Known skin or scalp conditions that may preclude attachment or interfere with the usage of the sound processor.
9. Known retro cochlear pathology and auditory processing disorders that may have an impact on the outcome of the investigation
10. Any other known condition that the investigator determines could interfere with compliance or investigation assessments.
11. Use of ototoxic drugs that could be harmful to the hearing, as judged by the investigator.
12. Subject that has received radiotherapy in the area of implantation or is planned for such radiotherapy or similar during the investigation period.
13. For bilateral asymmetric candidates, subject already treated with a bone-anchored hearing solution on the side with the best bone conduction thresholds
14. Known chronic or non-revisable vestibular or balance disorder
15. Known abnormally progressive hearing loss
16. For conductive and mixed losses: evidence that hearing loss is retro-cochlear or of central origin
17. Participation in another clinical investigation with pharmaceuticals and/or devices which might cause interference with investigation participation.
18. Use of active implantable or body worn device that for medical reasons cannot be removed or discontinued, such as implantable cardiac pacemakers, defibrillators, or neurostimulators.
19. Known need for frequent MRI investigations for follow-up of other diseases.
20. Any subject that according to the Declaration of Helsinki is deemed unsuitable for investigation enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Demonstrate that the Sentio system improves hearing on the implanted ear. | 3 months post-surgery
  Functional gain with Sentio, i.e. the difference between preoperative unaided and aided sound field thresholds on the implanted ear.
Demonstrate that the Sentio system provides patients with improved speech recognition on the implanted ear. | 3 months post-surgery
  Difference in speech recognition score in percent between pre-operative unaided condition and aided with Sentio, measured in quiet on the implanted ear.

SECONDARY OUTCOMES:
Thorough assessment of performance (functional gain, effective gain, speech recognition), satisfaction, usability, comfort and health-related quality of life. | 3-24 months post-surgery
  Sound field audiometry, speech testing in quiet and noise and patient reported outcomes on listed topics.

OTHER OUTCOMES:
Evaluate the safety profile of the Sentio system in terms of the occurrence of adverse events and serious adverse events related to the device. | 3 months post-surgery
  Tabulated adverse events and serious adverse events related to the device reported from surgery throughout the investigation reported at 3 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Myrthe Hol, MD, PhD, Principal Investigator — ENT Department, University Medical Center Groningen; Emmanuel Mylanus, MD, PhD, Principal Investigator — ENT Department, Radboud University Medical Center; Peter Monksfield, MD, PhD, Principal Investigator — ENT - University Hospitals Birmingham NHS, Foundation Trust; James Tysome, MD, PhD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust, Addenbrookes Hospital; Susan Arndt, MD, PhD, Principal Investigator — Universitätsklinikum Freiburg; Thomas Lenartz, MD, PhD, Study Director — HNO-Klinik Medizinische Hochschule Hannover
Locations (6):
- Germany (2):
  - Universitätsklinikum Freiburg Universitätsklinik für Hals,- Nasen und Ohrenheilkunde, Freiburg im Breisgau
  - HNO-Klinik Medizinische Hochschule Hanover, Hanover
- Netherlands (2):
  - ENT Department, University Medical Center Groningen, Groningen
  - ENT department Radboud University Medical Center (Radboud UMC), Nijmegen
- United Kingdom (2):
  - ENT - University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital Birmingham, Birmingham
  - Cambridge University Hospitals NHS Foundation Trust, Addenbrookes Hospital, Cambridge

IPD SHARING:
Plan to Share IPD: No